CLINICAL TRIAL: NCT05163912
Title: A Virtual Home Intervention to Promote Physical Activity Among Youth With Type 1 Diabetes
Brief Title: Virtual Physical Activity for Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Robert E. Leet and Clara Guthrie Patterson Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000030105; 852679 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2021-12-09; First posted 2021-12-20 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: Exercise; Adolescent; Video games; Self-management; Social support
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Virtual home intervention
  Interventions: Behavioral: Virtual home intervention

INTERVENTIONS:
Behavioral: Virtual home intervention — Group classes with active videogames and discussions

SUMMARY:
A virtual group of teens with type 1 diabetes, led by young adults with type 1 diabetes, will play active videogames and discuss activity and health. This study will evaluate the program for feasibility and user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age of 14-19 years
* Diagnosis of type 1 diabetes or other absolute insulin deficiency diabetes for ≥6 months
* Inadequate moderate-to-vigorous physical activity levels (defined as ≤3 days per week achieving ≥60min daily, which is ≤50% of the recommended 7 days per week)
* English literacy
* Own a continuous glucose monitor (Dexcom G4, G5, G6 [San Diego, CA], Abbott Freestyle Libre 2, 14-day [Chicago, IL], Medtronic Guardian 3, Enlite [Dublin, Ireland]) with enough supplies for 6 weeks (when available, we will provide these to those who do not own them, in which case they will be considered to meet this criteria).
* Access to television or computer with HDMI or USB port.
* Under regular care by a healthcare provider (defined as attending at least one appointment in the past year, plus access to verified 24hr phone number to reach the provider's team for insulin dose adjustments if assistance is needed)

Exclusion Criteria:

• A condition or disability besides type 1 diabetes that would preclude participation in group moderate-to-vigorous physical activity (e.g., cerebral palsy, current pregnancy)

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Adherence | 6 weeks
  Number of group classes attended
Acceptability | 6 weeks
  Score on a satisfaction survey that has been custom-designed for the components of this program. Scores range from 0 to 4. A higher score indicates greater satisfaction with the program.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mak SS, Nally LM, Montoya J, Marrero R, DeJonckheere M, Joiner KL, Nam S, Ash GI. An Exergames Program for Adolescents With Type 1 Diabetes: Qualitative Study of Acceptability. JMIR Diabetes. 2025 May 28;10:e65665. doi: 10.2196/65665. PMID 40238214